CLINICAL TRIAL: NCT06037356
Title: Prostatic Urethral Lift Versus Transurethral Resection of Prostate in Benign Prostatic Hyperplasia Patients With Urinary Retention
Brief Title: PUL vs TURP in BPH Patients With Urinary Retention
Acronym: PULTUR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Brian Ho, Associate Consultant, Queen Mary Hospital, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QMH PULTUR Study
Record Dates: First submitted 2023-04-26; First posted 2023-09-14 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: BPH With Urinary Obstruction
Keywords: BPH; Urinary retention; prostatic urethral lift; PUL; TURP
MeSH Terms: conditions — Urinary Retention | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Intervention Model Description: The study will be a prospective, non-inferiority randomized controlled trial with the aim of detecting a non-inferiority margin of 5%. Subjects will be randomized in a 1:1 ratio.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Prostatic Urethral Lift (Experimental): Prostatic urethral lift implants will be placed in patients under local anesthesia or monitored anesthetic care. The number of implants used will depend on intra-operative findings, ranging from 2 to 8 implants per patient.
  Interventions: Device: Prostatic Urethral Lift
- TURP (Active Comparator): Transurethral resection of prostate (TURP) will be performed under spinal or general anesthesia as per usual care.
  Interventions: Procedure: TURP

INTERVENTIONS:
Device: Prostatic Urethral Lift — Prostatic urethral lift uses permanent implants to retract the prostate lobes away from the prostate urethra to allow unobstructed passage of urine. These implants are made of Nitinol, non-absorbable monofilament suture material (Poly Ethylene Terephthalate), Stainless Steel
  Other Names: PUL; Urolift
  Arms: Prostatic Urethral Lift
Procedure: TURP — Using monopolar or bipolar loop diathermy via cystoscopy, excess prostate tissue is resected piecemeal to remove obstruction to the prostatic urethra due to BPH
  Other Names: Transurethral resection of prostate
  Arms: TURP

SUMMARY:
The study will be a prospective, randomized controlled trial comparing prostatic urethral lift (PUL) versus transurethral resection of prostate (TURP) in benign prostate hyperplasia (BPH) patients with urinary retention. The primary objective of this study is to compare the catheter-free rates of PUL vs TURP. Secondary objectives include comparison of complications rates, cost effectiveness, patient satisfactory, symptom scores, quality of life measures and urodynamic parameters.

DETAILED DESCRIPTION:
The study will be a prospective, non-inferiority randomized controlled trial with the aim of detecting a non-inferiority margin of 5%.

After the potential subject has been informed of the study and the potential risks, he will be screened for eligibility within a 4 week period. Assessment of eligibility will include questionnaires, blood tests, urine tests, uroflowmetry, flexible cystoscopy, transrectal ultrasound, and urodynamic study. Suitable subjects will then be randomized in a 1:1 ratio to the prostatic urethral lift (intervention group) and TURP (control group). Patients in the prostatic urethral lift will have the procedure performed under local anesthesia or monitored anesthetic care while TURP patients will be performed under spinal or general anesthesia. The subjects will have regular follow up 1 month, 3 months, 6 months, 1 year, 2 years, 3 years, 4 years, and 5 years post-operatively. Follow up assessments will include questionnaires, uroflowmetry, and occasional urodynamic study.

ELIGIBILITY:
Inclusion Criteria:

* Male patients
* age >40 years old
* urinary retention who failed trial without catheter

Exclusion Criteria:

* Inability to provide consent OR no guardians or relatives to help provide consent on patient's behalf
* Active urinary tract infection
* Previous surgical treatment for benign prostatic hyperplasia (i.e., TURP, prostatic urethral lift, etc.)
* Bladder stones
* Urethral strictures or bladder neck contractures
* Prostate size >100mL
* Solely obstructing median lobe
* Urinary retention not due to obstruction (i.e., Bladder outflow obstruction index <20 on urodynamic studies)
* Poor detrusor contractility (maximum detrusor pressure <20cmH2O during voiding phase)
* Anticoagulant or antiplatelet agents that cannot be stopped

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2035-05-30 (Estimated); Study Completion 2035-05-30 (Estimated)

PRIMARY OUTCOMES:
Catheter-free rates after prostatic urethral lift versus TURP in BPH patients with urinary retention | 1 year after intervention
  To determine how many patients will be catheter-free (defined as by the ability to void with a post-void residual urine <300mL) after intervention and remain catheter-free at 1 month, 3 months, and 1 year after intervention

SECONDARY OUTCOMES:
Compare complication rate of prostatic urethral lift versus TURP in BPH patients with urinary retention | 5 years
  To determine the percentage and severity of complications after each intervention (according to the Clavien-Dindo classification)
Cost effectiveness of prostatic urethral lift versus TURP in achieving catheter-free rates in BPH patients with urinary retention | 1 year
  To determine the cost required to achieve catheter free patients for each intervention (including hospitalization, anesthetic costs, equipment, consumables, etc)
Compare patient satisfaction by PGI-I questionnaire after prostatic urethral lift versus TURP | 1 year
  Using the Patient global impression of improvement (PGI-I) questionnaire to determine patient satisfaction after each intervention.
  * minimum score is 1, maximum score is 7
  * higher score means worse outcome
Compare patient reported symptom measures by IPSS questionnaire after prostatic urethral lift versus TURP | 1 year
  Using International prostate symptom score (IPSS) questionnaire to determine patient reported symptom measure after each intervention
  * minimal score: 0, maximum score is 35
  * higher score means worse outcome
Compare patient reported symptom measures by ISI questionnaire after prostatic urethral lift versus TURP | 1 year
  Using the Incontinence severity index (ISI) questionnaire to determine patient reported symptom measure after each intervention
  * minimum score: 1, maximum score: 12
  * higher score means worse outcome
Compare patient reported symptom measures by IIEF-5 questionnaire after prostatic urethral lift versus TURP | 1 year
  Using the International index of erectile function- 5 items (IIEF-5) questionnaire to determine patient reported symptom measure after each intervention
  * minimum score: 1, maximum score: 25
  * higher score means better outcome
Compare patient reported symptom measures by MSHQ-EjD short form questionnaire after prostatic urethral lift versus TURP | 1 year
  Using the Male Sexual Health Questionnaire for Ejaculatory Dysfunction (MSHQ-EjD) short form questionnaire to determine patient reported symptom measure after each intervention.
Compare patient reported quality of life by SF-12 questionnaire after prostatic urethral lift versus TURP | 1 year
  Using the Short Form 12 (SF-12) questionnaire to determine patient reported quality of life measures after each intervention
  * minimum score: 0, maximum score: 100
  * higher score means better outcome
Compare patient reported quality of life by derived SF-6D utility score after prostatic urethral lift versus TURP | 1 year
  Using the derived Short Form 6 Dimension (SF-6D) utility score questionnaire to determine patient reported quality of life measures after each intervention
  * minimum score: 0, maximum score 1.0
  * higher score means better outcome
Compare patient reported recovery by VAS after prostatic urethral lift versus TURP | 1 year
  Using the Visual analogue scale of quality of recovery to determine patient reported recovery after each intervention
  * minimum score: 0, maximum score 100
  * higher score means better outcome
Compare improvement bladder contractility index after prostatic urethral lift versus TURP | 5 year
  Pre- and post-intervention urodynamic will be performed to assess bladder contractility index as well as subsequent improvement and durability of above stated urodynamic parameter after each intervention
Compare improvement of Bladder outflow obstruction index after prostatic urethral lift versus TURP | 5 year
  Pre- and post-intervention urodynamic will be performed to assess bladder outflow obstruction index (BOOI) as well as subsequent improvement and durability of above stated urodynamic parameter after each intervention

CONTACTS AND LOCATIONS:
Overall Officials: Brian SH Ho, MBBS, Principal Investigator — Queen Mary Hospital, Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garraway WM, Collins GN, Lee RJ. High prevalence of benign prostatic hypertrophy in the community. Lancet. 1991 Aug 24;338(8765):469-71. doi: 10.1016/0140-6736(91)90543-x. PMID 1714529
- [Background] Jacobsen SJ, Jacobson DJ, Girman CJ, Roberts RO, Rhodes T, Guess HA, Lieber MM. Treatment for benign prostatic hyperplasia among community dwelling men: the Olmsted County study of urinary symptoms and health status. J Urol. 1999 Oct;162(4):1301-6. PMID 10492184
- [Background] Madersbacher S, Marberger M. Is transurethral resection of the prostate still justified? BJU Int. 1999 Feb;83(3):227-37. doi: 10.1046/j.1464-410x.1999.00908.x. No abstract available. PMID 10233485
- [Background] Mebust WK, Holtgrewe HL, Cockett AT, Peters PC. Transurethral prostatectomy: immediate and postoperative complications. a cooperative study of 13 participating institutions evaluating 3,885 patients. 1989. J Urol. 2002 Feb;167(2 Pt 2):999-1003; discussion 1004. No abstract available. PMID 11908420
- [Background] Neal DE. The National Prostatectomy Audit. Br J Urol. 1997 Apr;79 Suppl 2:69-75. doi: 10.1111/j.1464-410x.1997.tb16924.x. No abstract available. PMID 9126073
- [Background] Woo HH, Chin PT, McNicholas TA, Gill HS, Plante MK, Bruskewitz RC, Roehrborn CG. Safety and feasibility of the prostatic urethral lift: a novel, minimally invasive treatment for lower urinary tract symptoms (LUTS) secondary to benign prostatic hyperplasia (BPH). BJU Int. 2011 Jul;108(1):82-8. doi: 10.1111/j.1464-410X.2011.10342.x. Epub 2011 May 6. PMID 21554526
- [Background] Walsh LP. State of the art: Advanced techniques for prostatic urethral lift for the relief of prostate obstruction under local anesthesia. Can J Urol. 2017 Jun;24(3):8859-8864. PMID 28646943
- [Background] Eure G, Gange S, Walter P, Khan A, Chabert C, Mueller T, Cozzi P, Patel M, Freedman S, Chin P, Ochs S, Hirsh A, Trotter M, Grier D. Real-World Evidence of Prostatic Urethral Lift Confirms Pivotal Clinical Study Results: 2-Year Outcomes of a Retrospective Multicenter Study. J Endourol. 2019 Jul;33(7):576-584. doi: 10.1089/end.2019.0167. Epub 2019 Jun 25. PMID 31115257
- [Background] Roehrborn CG, Barkin J, Gange SN, Shore ND, Giddens JL, Bolton DM, Cowan BE, Cantwell AL, McVary KT, Te AE, Gholami SS, Moseley WG, Chin PT, Dowling WT, Freedman SJ, Incze PF, Coffield KS, Herron S, Rashid P, Rukstalis DB. Five year results of the prospective randomized controlled prostatic urethral L.I.F.T. study. Can J Urol. 2017 Jun;24(3):8802-8813. PMID 28646935
- [Background] McVary KT, Gange SN, Shore ND, Bolton DM, Cowan BE, Brown BT, Te AE, Chin PT, Rukstalis DB, Roehrborn CG; L.I.F.T. Study Investigators. Treatment of LUTS secondary to BPH while preserving sexual function: randomized controlled study of prostatic urethral lift. J Sex Med. 2014 Jan;11(1):279-87. doi: 10.1111/jsm.12333. Epub 2013 Sep 30. PMID 24119101
- [Background] Sievert KD, Schonthaler M, Berges R, Toomey P, Drager D, Herlemann A, Miller F, Wetterauer U, Volkmer B, Gratzke C, Amend B. Minimally invasive prostatic urethral lift (PUL) efficacious in TURP candidates: a multicenter German evaluation after 2 years. World J Urol. 2019 Jul;37(7):1353-1360. doi: 10.1007/s00345-018-2494-1. Epub 2018 Oct 3. PMID 30283994